CLINICAL TRIAL: NCT05324683
Title: "ILUMIEN-V - AERO"- All-comEr Registry of OCT (AERO) to Investigate the MLD-MAX Algorithm for OCT-guided-precision-PCI in Daily Routine
Brief Title: ILUMIEN-V - AERO: All-comEr Registry of OCT (AERO)
Status: Recruiting | Type: Observational
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: ILUMIEN-V - AERO V 1.2
Record Dates: First submitted 2022-04-06; First posted 2022-04-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study population (cohort): No study arms; one patient population will be observed.
  Interventions: Other: No intervention planned

INTERVENTIONS:
Other: No intervention planned — No intervention planned; study is observational

SUMMARY:
The study aims to assess contemporary practice in OCT use during routine interven-tional practice and to assess the impact of the MLD-MAX algorithm on real-world PCI in a large unselected European all-comer-study cohort.

DETAILED DESCRIPTION:
Angiography is the current standard method to guide PCI strategy in clinical practice. However, angiography has a number of well-described limitations, primarily through only providing an assessment of luminal dimensions without delineation of the burden of atheroma-tous disease. Angiography also provides suboptimal assessment of post PCI complications such as stent underexpansion or malapposi-tion, residual dissections or thrombus, and tissue prolapse. These limi-tations may be overcome in part by intravascular imaging (IVI), which allows tomographic, cross-sectional imaging of the vessel wall. Meta-analyses of randomized and registry studies of IVI-guided vs. angi-ography-guided PCI have suggested that IVI-guidance may improve clinical outcome following PCI.

Optical coherence tomography (OCT) provides high-resolution (10-20 μm) cross-sectional images of plaque microarchitecture, stent place-ment and size and strut coverage. Recently the MLD-MAX algorithm was developed to guide and stand-ardize coronary stent implantation based on sizing of the vessel at the proximal and distal reference using the EEL.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with evidence of myocardial ischemia (e.g. stable angi-na, silent ischemia, unstable angina, or acute myocardial infarc-tion) undergoing OCT-guided lesion evaluation (OCT-scan using the devices must be performed either to guide PCI (following the MLD-MAX-algorithm) or to investigate a coronary lesion for fur-ther clinical treatment)
* Written informed consent (defined as legally effective, docu-mented confirmation of a subject's (or their legally authorized representative or guardian) voluntary agreement to participate in a particular clinical study) to participate in this clinical inves-tigation

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with evidence of myocardial ischemia (e.g. stable angina, silent ischemia, unstable angina, or acute myocardial infarction) un-dergoing OCT-guided lesion evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Stent expansion: number of participants with optimal / acceptable / unacceptable stent expansion | At baseline
  Stent expansion is defined by the MSA achieved in the proximal and distal stented segments relative to their respective reference lumen areas. Stent expansion will be categorised as follows:
  Optimal stent expansion (y/n); acceptable stent expansion (y/n); unacceptable stent expansion (y/n); post-PCI stent expansion (%).

SECONDARY OUTCOMES:
Minimal Stent Area (MSA) | At baseline
  Imaging Outcome: minimal stent area as continuous measure; Final Post-PCI MSA (per target lesion basis) assessed by final-OCT after PCI; measured at an independent OCT core laboratory. Imaging-Outcome: Minimal-Stent-Area (MSA), continuous measure
Mean stent expansion | At baseline
  The mean stent area (stent volume/analyzed stent length) divided by the average of proximal and distal reference lumen areas x 100
Intra-stent plaque protrusion and thrombus: number of major and minor protusion area / stent area | At baseline
  Defined as a mass attached to the luminal surface or floating within the lumen, meeting the following criteria: Protrusion/thrombus is defined as any intraluminal mass protruding at least 0.2 mm within the luminal edge of a stent strut, and will be further classified as Major and Minor:
  * Major: Protrusion area/Stent area at site of tissue protrusion ≥10% and the minimal intra-stent flow area (MSA - protrusion area) is unacceptable (<90% of respective proximal or distal reference area
  * Minor: Protrusion area/Stent area at site of tissue protrusion is <10%, or is ≥10% but the minimal intraluminal flow area (MSA - protrusion area) is acceptable (≥90% of respective proximal or distal reference area
Number of participants with untreated reference segmant disease | At baseline
  Defined as focal disease with untreated MLA <4.5 mm2 within 5 mm from the proximal and/or distal stent edges. Sub-classified by the amount of untreated lipid plaque, divided into 3 grades: Low (≤90° of lipid arc), Medium (>90°-<180° of lipid arc) and High (≥180° of lipid arc).
Number of participants with major and minor edge dissections | At baseline
  Edge dissections will be tabulated as:
  * Major (%): ≥60 degrees of the circumference of the vessel at site of dissection and ≥3 mm in length
  * Minor (%): any visible edge dissection <60 degrees of the cir-cumference of the vessel or <3 mm in length
Number of participants with major and minor stent malapposition | At baseline
  Defined as frequency (%) of incompletely apposed stent struts (defined as stent struts clearly separated from the vessel wall (lumen bor-der/plaque surface) without any tissue behind the struts with a distance from the adjacent intima of ≥0.2 mm and not associated with any side branch). Malapposition will be further classified as:
  * Major: if associated with unacceptable stent expansion (as de-fined above)
  * Minor: if associated with acceptable stent expansion (as defined above) Stent Malapposition will be tabulated as: Major (%); Minor (%); All (Major and Minor) (%)
Number of participants with procedural complications | At baseline
  Defined as prolonged ST-segment elevation or depression (>30 minutes), cardiac arrest or need for defibrillation or cardioversion or hypotension/heart failure requiring mechanical or intravenous hemody-namic support or intubation or procedural death
Number of participants with adverse events | At 30 days follow-up
  Target lesion failure (TLF; cardiac death, TV-MI or ischemia-driven target lesion revascularization)
Number of participants with adverse events | At 6 months follow-up
  Target lesion failure (TLF; cardiac death, TV-MI or ischemia-driven target lesion revascularization)

CONTACTS AND LOCATIONS:
Overall Officials: David-Manuel Leistner, Prof Dr med, Principal Investigator — Universitätsklinikum Frankfurt - Med. Klinik 3 - Kardiologie; Thomas Johnson, Dr med, Principal Investigator — Bristol Heart Institute
Locations (1):
- Universitätsklinikum Frankfurt - Med. Klinik 3 - Kardiologie, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No